CLINICAL TRIAL: NCT06820567
Title: English Title of Research Project: Effects of Dapagliflozin on Inflammatory Markers, Erythropoiesis and Iron Metabolism in Patients with Type 2 Diabetes and CKD
Brief Title: Effects Dapagliflozin on Inflammatory Markers Erythropoiesis and Iron Metabolism in Patients with Type 2 Diabetes and CKD
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zeinab Khodary Saady Ali, residant doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: effect Dapagliflozin on CKD
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Diseases; Diabetes Type 2
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): type 2 diabetic patients with chronic kidney diseases will recive dapagliflozin
  Interventions: Drug: Dapagliflozin (DAPA)
- Group B (Placebo Comparator): type 2 diabetic patients with chronic kidney diseases will recive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin (DAPA) — patient will recive dapagliflozin for 24 week to improvement of eGFR on CKD patients
  Arms: Group A
Drug: Placebo — type 2 diabetic patients with chronic kidney diseases will recive placebo for 24 weeks
  Arms: Group B

SUMMARY:
the effect of Dapagliflozin on erythropoiesis, iron metabolism and inflammatory markers in CKD with Type 2 DM-Compare between effect of placebo and dapagliflozin on erythropoiesis, iron metabolism and inflammation markers in CKD with Type 2 DM.

DETAILED DESCRIPTION:
Type 2 diabetes is considered an important cause of chronic kidney diseases (CKD) ,in those patients the inflammation is the most assumed cause of the decrease in erythropoietin synthesis and abnormal iron metabolism leading to anemia (1_3).

Sodium glucose cotransporter 2 (SGLT2) inhibitors like Dapagliflozin are oral medications approved for type 2 diabetes. interestingly, during recent years, they have been promisingly considered as anew medications for cardiovascular and kidney diseases (4). Researchers suggested that SGLT 2 inhibitors play an important role in reducing CKD progression and renal failure with patients with type 2 DM based on the clinical outcomes and laboratory findings rather than completely understood mechanism (5_8)

Investigators reported that reduced transferrin saturation (TSAT), ferritin and hepcidin and circulating and urinary inflammatory mediators, including monocyte chemoattractant protein-1 (MCP -1 ) and interleukin-6 (IL-6) transiently increased EPO suggesting SGLT 2 inhibition may help iron utilization and promote erythropoiesis decreasing anemia ( 9-14)

Here we are studying the effects of the SGLT 2 inhibitor Dapagliflozin regarding markers of erythropoiesis, iron metabolism and inflammation in patients with Type 2 DM and CKD.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants were aged >18 years and diagnosed with Type 2 diabetes participants we required to have urinary albumin-creatinine ratio (UACR ) of 30_3500 mg /g ,eGFR of 20_ 80 ml/min/ 1.73 m , and HbA1c of 7.0 _ 11.0 % at screening

Exclusion Criteria:

type 1 diabetes, non-diabetes kidney disease and patient with HB < 9

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
GFR in CKD patients | 6 months
  Measure eGFR using ckd epi equation to detect the effect of dapagliflozin in improvement of GFR in CKD patients

CONTACTS AND LOCATIONS:
Overall Officials: Mai Mostafa, MD, Study Director — professor

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Koshino A, Neuen BL, Jongs N, Pollock C, Greasley PJ, Andersson EM, Hammarstedt A, Karlsson C, Langkilde AM, Wada T, Heerspink HJL. Effects of dapagliflozin and dapagliflozin-saxagliptin on erythropoiesis, iron and inflammation markers in patients with type 2 diabetes and chronic kidney disease: data from the DELIGHT trial. Cardiovasc Diabetol. 2023 Nov 28;22(1):330. doi: 10.1186/s12933-023-02027-8. PMID 38017482